CLINICAL TRIAL: NCT02355561
Title: An Open-Label, Randomized, Three-Period Crossover Study to Evaluate the Relative Oral Bioavailability and Food Effect of JNJ-54861911 Tablet (1x25mg) After Single Dose Administration in Healthy Elderly Subjects
Brief Title: A Crossover Study to Evaluate the Relative Oral Bioavailability and Food Effect After Single Dose Administration of JNJ-54861911 Tablet in Healthy Elderly Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR106621; 2014-004251-31 (EudraCT Number); 54861911ALZ1011 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Healthy
Keywords: Bioavailability; Healthy Participants; JNJ-54861911; Food Effect
MeSH Terms: interventions — atabecestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1 (ABC) (Experimental): Participants will receive Treatment A (single dose of JNJ-54861911 25 milligram [mg] formulation 1 [reference] under fasted conditions) in Period 1; followed by Treatment B (single oral dose of JNJ-54861911 25 mg formulation 2 [test] under fasted conditions) in Period 2; followed by Treatment C (single oral dose of JNJ-54861911 25 mg formulation 2 under fed conditions) in Period 3. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-54861911 (Treatment A); Drug: JNJ-54861911 (Treatment B); Drug: JNJ-54861911 (Treatment C)
- Sequence 2 (ACB) (Experimental): Participants will receive Treatment A in Period 1; followed by Treatment C in Period 2; followed by Treatment B in Period 3. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-54861911 (Treatment A); Drug: JNJ-54861911 (Treatment B); Drug: JNJ-54861911 (Treatment C)
- Sequence 3 (BAC) (Experimental): Participants will receive Treatment B in Period 1; followed by Treatment A in Period 2; followed by Treatment C in Period 3. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-54861911 (Treatment A); Drug: JNJ-54861911 (Treatment B); Drug: JNJ-54861911 (Treatment C)
- Sequence 4 (BCA) (Experimental): Participants will receive Treatment B in Period 1; followed by Treatment C in Period 2; followed by Treatment A in Period 3. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-54861911 (Treatment A); Drug: JNJ-54861911 (Treatment B); Drug: JNJ-54861911 (Treatment C)
- Sequence 5 (CAB) (Experimental): Participants will receive Treatment C in Period 1; followed by Treatment A in Period 2; followed by Treatment B in Period 3. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-54861911 (Treatment A); Drug: JNJ-54861911 (Treatment B); Drug: JNJ-54861911 (Treatment C)
- Sequence 6 (CBA) (Experimental): Participants will receive Treatment C in Period 1; followed by Treatment B in Period 2; followed by Treatment A in Period 3. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-54861911 (Treatment A); Drug: JNJ-54861911 (Treatment B); Drug: JNJ-54861911 (Treatment C)

INTERVENTIONS:
Drug: JNJ-54861911 (Treatment A) — Participants will receive a single oral 25 mg formulation 1 of JNJ-54861911 tablet as Treatment A under fasted conditions in one of the treatment periods.
Drug: JNJ-54861911 (Treatment B) — Participants will receive a single oral 25 mg formulation 2 of JNJ-54861911 tablet as Treatment B under fasted conditions in one of the treatment periods.
Drug: JNJ-54861911 (Treatment C) — Participants will receive a single oral 25 mg formulation 2 of JNJ-54861911 tablet as Treatment C under fed conditions in one of the treatment periods.

SUMMARY:
The purpose of this study is to assess the effect of a high-fat/high-caloric breakfast on the rate and extent of absorption of the single oral dose of 25 mg JNJ-54861911 test formulation in healthy elderly participants.

DETAILED DESCRIPTION:
This is a randomized (study medication assigned to participants by chance), open-label (all people know the identity of the intervention), 3-treatment, 3-period, 6-sequence crossover (participants may receive different interventions sequentially during the trial), and single-center study of JNJ-54861911. The duration of study will be approximately of 7 weeks per participant. The study consists of 3 parts: Screening (that is, 21 days before study commences on Day 1); Open-label Treatment (consists of 3 single-dose treatments, either JNJ-54861911 formulation 1 [reference] or JNJ-54861911 formulation 2 [test] under fed or fasted condition), in subsequent 3-treatment periods, each separated with washout period of 7 days); and End-of-Study (up-to 14 days after last study drug administration). All the eligible participants will be randomly assigned to 1 of the 6 treatment sequences. In fasted conditions, study drug will be administered following a 10-hour overnight fast. In fed conditions, participants will also fast from food for 10 hours, but will consume a high fat/high calorie breakfast within a 30-minute period. Study drug will be administered 30 minutes after the start of breakfast. Participants will not be allowed to have food until 4 hours of drug administration. Blood samples will be collected for evaluation of pharmacokinetics at pre-dose and post-dose of study treatment. Relative bioavailability of two formulations of JNJ-54861911 (test and reference) will be evaluated primarily. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a body mass index (BMI) between 18 and 30 Kilogram (kg)/Meter (m)^2, inclusive (BMI = weight/height^2)
* Participant must be healthy for their age group with or without medication on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at Screening and admission. Minor deviations in ECG, which are not considered to be of clinical significance to the investigator, are acceptable
* Participants must be healthy on the basis of clinical laboratory tests performed at Screening. If the results of the serum chemistry panel [including liver enzymes], hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* Before randomization, a woman must be not of childbearing potential: postmenopausal (greater than or equal to [≥] 55 years of age with amenorrhea for at least 12 months; permanently sterilized [e.g., tubal occlusion, hysterectomy, bilateral salpingectomy]); or otherwise be incapable of pregnancy. In case of questionable status qualified personal of the sponsor should be consulted to decide on the potential for inclusion of the participant
* Men who are sexually active with a woman of childbearing potential and have not had a vasectomy must agree to use a barrier method of birth control e.g., either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the study and for 90 days after receiving the last dose of study drug. In addition, their female partners should also use an appropriate method of birth control for at least the same duration. Effective methods of contraception include prescription oral contraceptives, contraceptive injections, intrauterine device, double barrier method, contraceptive patch

Exclusion Criteria:

* Participant has clinically significant abnormal findings in physical exam, vital signs or 12-lead ECG incl. QTcF greater than (>) 450 milliseconds (ms) for males and females, Left Bundle Branch Block, Atrioventricular (AV) Block second degree or higher, permanent pacemaker or implantable cardioverter defibrillator (ICD) at Screening or admission, which in the opinion of the investigator are not appropriate and reasonable for the population under study
* Participant has a history of or current significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematological disease, lipid abnormalities, bronchospastic respiratory disease, diabetes mellitus, thyroid disease, Parkinson's disease, infection, or any other illness that the Investigator considers should exclude the participant
* Participant has a history of or current renal [Estimated glomerular filtration rate (eGFR) less than (<) 60 based on Modification of diet in renal diseases (MDRD) formula] or hepatic insufficiency
* Participant has a history of epilepsy or fits or unexplained black-outs other than vasovagal collapse
* Participant has a history of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease, or tests positive for HBsAg or anti-HCV at Screening

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of JNJ-54861911 | Pre-dose; 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post-dose on Day 1 of each period
  The Cmax is the maximum observed plasma concentration of JNJ-54861911.
Time to Reach the Maximum Plasma Concentration (Tmax) of JNJ-54861911 | Pre-dose; 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post-dose on Day 1 of each period
  The Tmax is the time to reach the maximum observed plasma concentration of JNJ-54861911.
Area Under the Plasma Concentration-Time Curve From 0 to t Hours (AUC[0-t]) Post Dose of JNJ-54861911 | Pre-dose; 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post-dose on Day 1 of each period
  The AUC (0-t) calculated by trapezoidal summation [time t is the time of the last quantifiable concentration (C[last])].
Area Under the Plasma Concentration-Time Curve From 0 to 24 Hours (AUC[0-24]) Post Dose of JNJ-54861911 | Pre-dose; 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post-dose on Day 1 of each period
  The AUC (0-24hrs) is the area under the plasma concentration-time curve from 0 to 24 hours post dosing.
Area Under the Plasma Concentration-Time Curve From 0 to Infinite Time (AUC[0-infinity]) Post Dose of JNJ-54861911 | Pre-dose; 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post-dose on Day 1 of each period
  The AUC (0-infinity) is the area under the plasma JNJ-54861911concentration-time curve from time 0 to infinite time, calculated as the sum of AUC (0-last) and C(last)/lambda(z), in which AUC(0-last) is area under the plasma JNJ-54861911 concentration-time curve from time zero to time of the last quantifiable concentration, C(last) is the last observed quantifiable concentration and lambda(z) is elimination rate constant.
Elimination Rate Constant (Lambda [z]) of JNJ-54861911 | Pre-dose; 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post-dose on Day 1 of each period
  The Lambda (z) determined by linear regression of the terminal points of the ln-linear plasma concentration-time curve.
Terminal Half-life (t[1/2]) of JNJ-54861911 | Pre-dose; 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post-dose on Day 1 of each period
  The t(1/2) is defined as 0.693/Lambda (z).
Relative Bioavailability (F[rel]) of JNJ-54861911 | Pre-dose; 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post-dose on Day 1 of each period
  Relative bioavailability, calculated as individual Cmax and AUC treatment ratios (for the comparison of food effect).

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious AEs | Screening up to follow-up (7 to 14 days after last dose administration)
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium